CLINICAL TRIAL: NCT05612867
Title: High Dose Intravenous Versus Low Dose Oral Vitamin C in Burn Care: Potential Protective Effects in the Severely Burned: A Retrospective Cohort Study
Brief Title: Low Dose Vitamin C in Burns >20% Compared to Previous Studies With High Dose Vitamin C
Status: Completed | Type: Observational
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-49
Record Dates: First submitted 2022-10-26; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Burns; Ascorbic Acid Deficiency; Burn Shock; Burn Degree Second; Burn Degree Third; Fluid and Electrolyte Imbalance
MeSH Terms: conditions — Burns; Ascorbic Acid Deficiency | interventions — Ascorbic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PO Vitamin C: Patients who got PO vitamin C
  Interventions: Dietary Supplement: Vitamin C
- IV Vitamin C: Patients who got IV vitamin C
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin C — Due to clinical research supporting high dose vitamin C, the institution's surgical intensivists started utilizing a high IV vitamin C dose in higher total body surface area burns while continuing to use the standard PO vitamin C dose of 500 mg to 1,000 mg daily on patients with lower total body surface area burns. Looking at the initial 72 hours, patients with smaller burns were given 2,500 mg PO vitamin C and larger total body surface area burns were given 15,000 mg IV vitamin C.

SUMMARY:
Burn injury is marked by a large release of inflammatory mediators which disrupt the normal capillary barrier and cause a rapid shift of intravascular fluid into interstitial spaces, ultimately leading to shock and death. As such, adequate fluid management and resuscitation is critical for burn patients to prevent further cellular injury. Technologies and medical options such as cardiac output monitoring along with early tube feeding and vitamin C administration have developed slowly over the years. Effective management of the Systemic Inflammatory Response Syndrome response and metabolic derangement is crucial for the survival of burn patients. In particular, vitamin C administration has shown to significantly decreases early post-burn lipid peroxidation, reduce microvascular leak of fluid by preventing endothelial dysfunction, and decreases edema formation in burned tissue. Vitamin C is a cheap and widely available antioxidant which has been shown to significantly effective in positively impacting clinical outcomes in burn resuscitation. We aim to evaluate the efficacy of vitamin C in burns greater than 20% total body surface area on clinical outcomes such as length of hospital stay, total fluid requirements, and mortality.

DETAILED DESCRIPTION:
Burn injury is marked by a large release of inflammatory mediators which disrupt the normal capillary barrier and cause a rapid shift of intravascular fluid into interstitial spaces, ultimately leading to shock and death. As such, adequate fluid management and resuscitation is critical for burn patients to prevent further cellular injury. Technologies and medical options such as cardiac output monitoring along with early tube feeding and vitamin C administration have developed slowly over the years. Effective management of the systemic inflammatory response syndrome response and metabolic derangement is crucial for the survival of burn patients. In particular, vitamin C administration has shown to significantly decreases early post-burn lipid peroxidation, reduce microvascular leak of fluid by preventing endothelial dysfunction, and decreases edema formation in burned tissue.

Vitamin C is a cheap and widely available antioxidant which has been shown to significantly effective in positively impacting clinical outcomes in burn resuscitation. While vitamin C is a regular part of burn resuscitation, there is no consensus on the most effective dose when considering impacting mortality, fluid resuscitation requirement, and other various clinical outcomes. Defining clinically efficacious minimal dosage of vitamin C can assist surgeons to better guide care for patients requiring burn resuscitation.

In this study, we aim to evaluate the efficacy of vitamin C in burns greater than 20% total body surface area on various clinical outcomes through a retrospective chart review of burn patients. Through this retrospective chart review, we aim to arrive at a better-defined vitamin C dose to achieve positive clinically significant outcomes.

ELIGIBILITY:
Inclusion Criteria:

All patients presenting to Arrowhead Regional Medical Center Emergency Department with International Classification of Diseases-10 codes of :

i. T31.2 Burns involving 20-29% of body surface ii. T31.3 Burns involving 30-39% of body surface iii. T31.4 Burns involving 40-49% of body surface iv. T31.5 Burns involving 50-59% of body surface v. T31.6 Burns involving 60-69% of body surface vi. T31.7 Burns involving 70-79% of body surface vii. T31.8 Burns involving 80-89% of body surface viii. T31.9 Burns involving 90% or more of body surface ix. T30.2 Burn of second degree, body region unspecified x. T30.3 Burn of third degree, body region unspecified

Exclusion Criteria:

* Total Body Surface Area Burns under 20%.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To evaluate PO vitamin C in burns of greater than 20% total body surface area compared to previous published studies utilizing high dose vitamin C in patients older than 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 hours
  Survival within the first 28 days
Infection rate | 180 days
  The time frame of any clinically documented infections and when they occurred
Ventilator days | 180 days
  The total duration of time a patient spends intubated on a ventilator while in the hospital. The initial intubation will be the only intubation considered
Fluid Requirement | 72 hours
  Total fluid requirements in first 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Aldin Malkoc, MD, Study Chair — Arrowhead Regional Medical Center; David T Wong, MD, Principal Investigator — Arrowhead Regional Medical Center
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanaka H, Matsuda H, Shimazaki S, Hanumadass M, Matsuda T. Reduced resuscitation fluid volume for second-degree burns with delayed initiation of ascorbic acid therapy. Arch Surg. 1997 Feb;132(2):158-61. doi: 10.1001/archsurg.1997.01430260056011. PMID 9041919
- [Background] Rock CL, Dechert RE, Khilnani R, Parker RS, Rodriguez JL. Carotenoids and antioxidant vitamins in patients after burn injury. J Burn Care Rehabil. 1997 May-Jun;18(3):269-78; discussion 268. doi: 10.1097/00004630-199705000-00018. PMID 9169953
- [Background] May JM. How does ascorbic acid prevent endothelial dysfunction? Free Radic Biol Med. 2000 May 1;28(9):1421-9. doi: 10.1016/s0891-5849(00)00269-0. PMID 10924860
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Barbosa E, Faintuch J, Machado Moreira EA, Goncalves da Silva VR, Lopes Pereima MJ, Martins Fagundes RL, Filho DW. Supplementation of vitamin E, vitamin C, and zinc attenuates oxidative stress in burned children: a randomized, double-blind, placebo-controlled pilot study. J Burn Care Res. 2009 Sep-Oct;30(5):859-66. doi: 10.1097/BCR.0b013e3181b487a8. PMID 19692922
- [Background] Wang Y, Lin H, Lin BW, Lin JD. Effects of different ascorbic acid doses on the mortality of critically ill patients: a meta-analysis. Ann Intensive Care. 2019 May 20;9(1):58. doi: 10.1186/s13613-019-0532-9. PMID 31111241
- [Result] Matsuda T, Tanaka H, Yuasa H, Forrest R, Matsuda H, Hanumadass M, Reyes H. The effects of high-dose vitamin C therapy on postburn lipid peroxidation. J Burn Care Rehabil. 1993 Nov-Dec;14(6):624-9. doi: 10.1097/00004630-199311000-00007. PMID 8300697